CLINICAL TRIAL: NCT01466777
Title: Robotic-assisted vs. Traditional Laparoscopic Surgery in Treatment of Endometrial Cancer Patients
Brief Title: Endometrial Cancer and Robotic-assisted Versus Traditional Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Minna Mäenpää, Principal Investigator, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R10081
Record Dates: First submitted 2011-08-18; First posted 2011-11-08 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Endometrium Cancer
Keywords: Endometrium cancer; Robotic-assisted laparoscopy; Traditional laparoscopy; Laparoscopic surgery; Treatment; Operation time; Bleeding; Complications; Conversions; Pelvic lymph node
MeSH Terms: conditions — Endometrial Neoplasms; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional laparoscopic surgery type (Active Comparator)
  Interventions: Procedure: Traditional surgery type
- Robotic assisted operation type (Experimental)
  Interventions: Procedure: Robotic assisted laparoscopic surgery

INTERVENTIONS:
Procedure: Traditional surgery type — Traditional laparoscopic surgery for endometrial cancer
  Arms: traditional laparoscopic surgery type
Procedure: Robotic assisted laparoscopic surgery — Robotic assisted laparoscopic surgery for endometrial cancer
  Arms: Robotic assisted operation type

SUMMARY:
The aim of this study is to compare the robotic-assisted laparoscopic surgery to the traditional laparoscopic surgery in endometrial cancer patients.

The study is prospective and the patients are randomised into two groups of 50 patients each. Randomisation is done with Minim-programme and patients age and Body mass index are taken into account.

The primary endpoint is the operation time. The number of patients in this study is based on the non-inferiority design. Presumption is that the operation time in robotic-assisted laparoscopy will be 25% longer.

Secondary endpoints include:

1. bleeding
2. complications
3. conversions
4. number of pelvic lymph nodes

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer operations, which means hysterectomy, bilateral salphingo-oophorectomy and pelvic lymphadenectomy
* Gr 1 and 2 differentiation type

Exclusion Criteria:

* The operation cannot be made with an laparoscopy operation
* Age more than 85 years or young under 30 years patient

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
the operation time | From the beginning of first wound incision to the closure of the wounds, an expected average of 3 hours

SECONDARY OUTCOMES:
bleeding | Duration of hospital stay, an expected average of 5 weeks
Number of participants with adverse events | Duration of hospital stay, an expected average of 5 weeks
Pain | Duration of hospital stay, an expected average of 5 weeks
  visual analogue scale
pelvic lymph node volumes | Duration of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, P.O.Box 2000, Finland

REFERENCES:
- [Derived] Vuorinen RK, Maenpaa MM, Nieminen K, Tomas EI, Luukkaala TH, Auvinen A, Maenpaa JU. Costs of Robotic-Assisted Versus Traditional Laparoscopy in Endometrial Cancer. Int J Gynecol Cancer. 2017 Oct;27(8):1788-1793. doi: 10.1097/IGC.0000000000001073. PMID 28937446